CLINICAL TRIAL: NCT06119919
Title: Cardiac Injury and it's Relation to Convulsive Status Epilepticus in Children
Brief Title: Cardiac Injury With Convulsive Status Epilepticus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Christin Emad Ragheb, 71515,Assiut, Assiut University
Other Study IDs: Cardiac injury and epilepsy
Record Dates: First submitted 2023-10-27; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Convulsive Status EPILEPTICUS
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Determine the impact of cardiac injury on clinical profile, cardiac evaluation and outcome in patients hospitalized with convulsive status epilepticus (CSE).
2. Analyze the frequency of cardiac rhythm and conduction abnormalities related to seizures and determine risk factors and associated clinical characteristics.
3. Analyse ECG abnormalities and changes in HR in epileptic seizures since such disturbances might be a factor in SUDEP
4. Assessment of levels of cardiac enzymes in patients with status epilepticus

DETAILED DESCRIPTION:
* Convulsive status epilepticus (CSE) is the most common life- threatening pediatric neurological emergency, with high morbidity and mortality rates . Previously, status epilepticus was defined as a seizure lasting more than 30 min . However, more recently, status epilepticus is considered if a patient has continuous seizure activity for 5 min or recurrent seizures without regaining consciousness level in between .
* Cardiac injury in CSE is associated with a combination of excessive catecholamine release, sympathetic overflow, and subsequent neurogenic myocardial stunning, resulting in subtle structural and functional myocardial damage with a high incidence of arrhythmia, stress-related cardiomyopathy, and heart failure moreover, cardiac injury may be iatrogenic due to intravenous fluid overload and cardio-depressive effects of anti-seizure medications (ASMs). Most of the SE-induced deaths occurring within 30 days following seizure activity are attributed to lethal cardiac arrhythmia, pulmonary edema, hypotension, and circulatory collapse
* Cardiac injury was defined as one or more of the following: (a) cardiac troponin ≥ 99th percentile , corrected for age and sex and (b) new- onset ECG changes categorized into ischemic changes, conduction abnormalities, or arrhythmias . (c) Left ventricular systolic or diastolic dysfunction, which is defined as follows: systolic dysfunction if EF < 56% and/or FS < 28% , diastolic dysfunction is defined and classified according to the recommendations of the American Society of Echocardiography and the European Association of Cardiovascular Imaging
* Changes in cardiac function in epilepsy imply an activation of the central autonomic network. In patients with seizures, epileptic discharges are thought to propagate to the central autonomic network and change or disturb normal autonomic control of vital cardiac functions. This activation of central autonomic nervous system is thought to be responsible for the peri-ictal autonomic cardiac symptoms observed in epilepsy patients. The importance of these autonomic features in the pathophysiology of epilepsy and its complications has become more clear in the last years.
* Conduction disorders seem to be common during seizures in intractable epilepsy could demonstrate the presence of arrhythmias or conduction disorders in seizures, particularly if these are prolonged or generalized. They include atrial fibrillation, supraventricular tachycardia and atrial and ventricular premature depolarisation. EKG changes, including T-wave inversion and ST-depression, were more frequent and potentially more dangerous in patients with generalized seizures.
* excessive autonomic stimulation may result in cardiac arrhythmias. But repetitive autonomic stimulation can also lead to structural damage to the heart. This increases the susceptibility to cardiac arrhythmias or ischemia. Myocardial fibrosis has already been found . Patients with uncomplicated seizures do not seem to have postictal troponin elevation, but signs of ischemia on ECG and elevated cardiac enzymes in epileptic patients suggest secondary cardiac damage could show presence of elevated Brain Natriuretic Peptide " BNP "and Creatine kinase Myocardial Band "CK-MB" in patients with seizures, the first evidence of subtle cardiac dysfunction in epilepsy patients.
* Cardiovascular-specific biomarkers have been identified as the most accurate indicators of myocardial infarction. Cardiovascular troponin-I (cTnI), in particular, is extremely selective for myocardial muscular tissue injury and is never produced following skeletal muscle injury .
* Patients with longlasting and multiple seizures seem to be prone to chronic dysfunction of autonomic cardiac control. In patients with newly diagnosed (median time 27 months) and untreated epilepsy, no difference was found in heart rate variability studied well controlled patients and refractory patients and could show with a series of autonomic tests that higher vasomotor tone, higher sympathetic tone, lower parasympathetic tone and reactivity was found in the group of refractory epilepsy patients. The observed dysautonomia could be a predisposing factor to SUDEP -sudden unexpected death in epilepsy. could demonstrate altered cardiovagal control in patients with chronic epilepsy.

ELIGIBILITY:
Inclusion Criteria:

1. children aged 1 month to 16 years presented with Convulsions
2. convulsions lasts more than 5 minutes or recurrent seizures without regaining consciousness in-between

Exclusion Criteria:

1. Patients with hepatic diseases
2. patients with chronic renal illness
3. patients with endocrinal diseases
4. patients with musculoskeletal abnormalities
5. children with sepsis
6. congenital heart disease, myocarditis, myocardial disease, or arrhythmias; and children who survived cardiac surgery

Ages: 1 Month to 16 Years | Sex: All
Age Groups: Child
Study Population: all children admitted in Assiut University Hospitals Pediatrics department from 1 month to 16 years with convulsive status epilepticus
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
cardiac injury and convulsive status epilepticus | baseline
  Determine the impact of cardiac injury on clinical profile and outcome in patients with convulsive status epilepticus
Cardiac injury and convulsive status epilepticus | Baseline
  Analyze the frequency of cardiac rhythm and conduction abnormalities
Cardiac injury and convulsive status epilepticus | Baseline
  Analyze ECG abnormalities and heart rate changes
Cardiac injury and convulsive status epilepticus | Baseline
  Assessment of levels of cardiac enzymes in patients with status epilepticus

REFERENCES:
- [Background] Fogarasi A, Janszky J, Tuxhorn I. Autonomic symptoms during childhood partial epileptic seizures. Epilepsia. 2006 Mar;47(3):584-8. doi: 10.1111/j.1528-1167.2006.00472.x. PMID 16529626
- [Background] Janszky J, Fogarasi A, Toth V, Magalova V, Gyimesi C, Kovacs N, Schulz R, Ebner A. Peri-ictal vegetative symptoms in temporal lobe epilepsy. Epilepsy Behav. 2007 Aug;11(1):125-9. doi: 10.1016/j.yebeh.2007.04.015. Epub 2007 Jun 20. PMID 17584534
- [Background] Widdess-Walsh P, Kotagal P, Jeha L, Wu G, Burgess R. Multiple auras: clinical significance and pathophysiology. Neurology. 2007 Aug 21;69(8):755-61. doi: 10.1212/01.wnl.0000267650.50269.5d. PMID 17709707
- [Background] Baumgartner C, Lurger S, Leutmezer F. Autonomic symptoms during epileptic seizures. Epileptic Disord. 2001 Sep;3(3):103-16. PMID 11679301
- [Background] Nei M, Ho RT, Sperling MR. EKG abnormalities during partial seizures in refractory epilepsy. Epilepsia. 2000 May;41(5):542-8. doi: 10.1111/j.1528-1157.2000.tb00207.x. PMID 10802759
- [Background] Natelson BH, Suarez RV, Terrence CF, Turizo R. Patients with epilepsy who die suddenly have cardiac disease. Arch Neurol. 1998 Jun;55(6):857-60. doi: 10.1001/archneur.55.6.857. PMID 9626779
- [Background] Woodruff BK, Britton JW, Tigaran S, Cascino GD, Burritt MF, McConnell JP, Ravkilde J, Molgaard H, Andreasen F, Dam M, Jaffe AS. Cardiac troponin levels following monitored epileptic seizures. Neurology. 2003 May 27;60(10):1690-2. doi: 10.1212/01.wnl.0000065881.46964.4f. PMID 12771269
- [Background] Tigaran S, Molgaard H, McClelland R, Dam M, Jaffe AS. Evidence of cardiac ischemia during seizures in drug refractory epilepsy patients. Neurology. 2003 Feb 11;60(3):492-5. doi: 10.1212/01.wnl.0000042090.13247.48. PMID 12578934
- [Background] Chin RF, Neville BG, Peckham C, Bedford H, Wade A, Scott RC; NLSTEPSS Collaborative Group. Incidence, cause, and short-term outcome of convulsive status epilepticus in childhood: prospective population-based study. Lancet. 2006 Jul 15;368(9531):222-9. doi: 10.1016/S0140-6736(06)69043-0. PMID 16844492
- [Background] Mitchell WG. Status epilepticus and acute serial seizures in children. J Child Neurol. 2002 Jan;17 Suppl 1:S36-43. doi: 10.1177/08830738020170010501. PMID 11918461